CLINICAL TRIAL: NCT04270877
Title: Fibromyalgia and Naltrexone: The FINAL Study
Acronym: FINAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Karin Bruun Plesner, Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18021; 2019-000702-30 (EudraCT Number); R177-A6158 (Other Grant/Funding Number: The Danish Reumatism Association); A3650 (Other Grant/Funding Number: The OUH PhD Committee for Operating Costs); 21-10-0037 (Other Grant/Funding Number: Aase and Ejnar Danielsens fund)
Record Dates: First submitted 2020-01-30; First posted 2020-02-17 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: A parallel randomized (1:1) double blind, placebo-controlled superior trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naltrexone (Experimental): Low Dose Naltrexone (LDN) is administered for 12 weeks, including a titration phase of 4 weeks.
  Participants will be titrated up to 6 mg following a dose escalation scheme: Initial dosage of 1.5 mg daily, escalated every seventh day by 1.5 mg up to 6 mg at week 4. Dose escalation will be based on safety and tolerability, and if dose escalation is not feasible, delayed increments are allowed. After end of titration (week 4) the subjects will be maintained at the highest tolerated dose level for the last 8 weeks of the treatment period. Subjects are not allowed to change dose during the last 8 weeks of the treatment period.
  The medicine is taken orally as tablets once daily in the evening.
  Interventions: Drug: Naltrexone Pill
- Placebo (Placebo Comparator): LDN-placebo is administered for 12 weeks, including a titration phase of 4 weeks.
  Participants will be titrated up to 6 mg following a dose escalation scheme: Initial dosage of 1.5 mg daily, escalated every seventh day by 1.5 mg up to 6 mg at week 4. Dose escalation will be based on safety and tolerability, and if dose escalation is not feasible, delayed increments are allowed. After end of titration (week 4) the subjects will be maintained at the highest tolerated dose level for the last 8 weeks of the treatment period. Subjects are not allowed to change dose during the last 8 weeks of the treatment period.
  The medicine is taken orally as tablets (similar in size, shape and taste to the active medication), once daily in the evening.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Naltrexone Pill — Treatment with LDN for 12 weeks, including af titration phase of 4 weeks. Initial dosage of 1.5 mg, dose is increased by 1.5 mg every 7th day to 6 mg at week 4. Dosing is increased based on safety and tolerability and delayed increments are allowed. The participants are maintained on the highest tolerable dose for the last 8 weeks of the treatment period.
  Other Names: LDN
  Arms: Naltrexone
Drug: Placebo oral tablet — Treatment with LDN-placebo for 12 weeks, including af titration phase of 4 weeks. Initial dosage of 1.5 mg, dose is increased by 1.5 mg every 7th day to 6 mg at week 4. Dosing is increased based on safety and tolerability and delayed increments are allowed. The participants are maintained on the highest tolerable dose for the last 8 weeks of the treatment period.
  Other Names: LDN-placebo
  Arms: Placebo

SUMMARY:
This study evaluates the effect of low dose naltrexone (LDN) on pain in women with fibromyalgia (FM). The study is designed as a parallel randomized (1:1) double blind, placebo-controlled superiority trial. Half of the participants will receive treatment with LDN while the other half will receive treatment with placebo.

DETAILED DESCRIPTION:
Low dose naltrexone (LDN) is used widely as off label treatment in patients with fibromyalgia, despite the lack of larger randomized controlled trials (RCT) supporting an effect.

LDN has antagonistic effect on both opioid receptors and on toll-like receptors in glia cells. Mediated via those receptors, LDN can potentially reduce neuroinflammation and induce homeostasis in the endorphin system in patients with fibromyalgia.

The aim of the trial is to investigate whether treatment with LDN has a superior effect compared to placebo on pain among female patients with fibromyalgia, evaluated after 12 weeks of treatment. The study is also exploring secondary aims regarding a possible improvement of other fibromyalgia core symptoms and a possible improvement of global assessment, daily functioning and health-related quality of life. Among the exploratory secondary objectives are changes in muscle exhaustion, physical fitness, pain sensitivity, inhibition of pain, augmentation of pain, and pro-inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-64 years
* Understands and writes Danish
* Fulfills the American College of Rheumatology 1990 criteria for fibromyalgia
* A minimum score of 4 in self-reported average pain during the last 7 days on a 0-10 numeric rating scale at baseline
* All fertile women have to use safe anti conception (Spiral, birth control pills, contraceptive patch, contraceptive vaginal ring or gestagen injections) for 3 weeks before and 1 week after the trial. If the patients' normal lifestyle includes sexual abstinence, they do not have to use anti conception. Instead they can give an oral informed consent, that they will be sexually abstinent during the trial. A woman is considered non-fertile if she is sterilized, hysterectomized, bilateral oophorectomized or is postmenopausal. A woman is considered postmenopausal when vaginal bleeding has been absent for 1 year and is confirmed by measurement of follicle-stimulating hormone.

Exclusion Criteria:

* Known allergy against naltrexonehydroclorid
* Pregnancy or breastfeeding. A negative pregnancy test has to be available for all fertile subjects at baseline
* Use of opioids or NSAIDs during the 4 weeks before inclusion in the trial
* Abuse of alcohol or other substances
* Inflammatory rheumatic diseases
* Demyelinating diseases
* Active cancer
* Liver dysfunction
* Kidney dysfunction
* Psychotic diseases
* History of suicide attempts
* Suicide ideation - evaluated using Patient Health Questionnaire-9 (Item 9 has to be answered "never")

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
Average pain during the last 7 days | Change from baseline when assessed after 12 weeks of treatment with LDN or LDN-placebo
  Assessed by asking the participants about the level of average pain during the last 7 days on a 11 point rating scale, ranging from 0-10 (0 = "no pain" and 10 = "unbearable pain") using the first item from the symptom part of the Fibromyalgia Impact Questionnaire Revised. A lower score indicates lower severity.

SECONDARY OUTCOMES:
Global assessment | Change in overall fibromyalgia symptoms from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Measured by Patient Global Impression of Change on a 1-7 Verbal Rating Scale. The participants are asked how they rate their overall fibromyalgia symptoms after 4, 8 and 12 weeks of treatment compared with before treatment. A score of 4 indicates "no change", a score of 1 is characterized by "a lot worse" and a score of 7 is characterized by "a lot better." A higher score indicates higher degree of improvement.
Impact of fibromyalgia | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Measured by the Fibromyalgia Impact Questionnaire Revised (FIQR) total score. The FIQR asks patients to rate how difficult it is to perform a list of 9 common activities over the previous 7 days on an 11 point scale, ranging from 0-10 (0 = "no difficulty" and 10 = "very difficult"). The FIQR then asks patients to indicate how often their fibromyalgia impacts their quality of life over the last 7 days on an 11 point scale, ranging from 1-10 (0 = "never" and 10 = "always"). Finally, the FIQR asks patients to assess the severity of 10 different symptoms on an 11 point scale, ranging from 0-10 (0 = "no symptoms" and 10 = "extreme symptoms"). These three sub-scales are summed to represent an overall FIQR score. A lower score indicates lower severity.
Pain distribution | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Assessed by the Widespread Pain Index (WPI) from The American College of Rheumatology 2016 revised criteria for fibromyalgia (ACR-2016). The body is divided into 19 body parts and number of pain full body parts during the last 7 days is counted, giving rise to the WPI. A lower score indicates lower spreading of pain.
Level of pain | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Assessed by the Fibromyalgia Impact Questionnaire Revised "level of pain" question, asking the participants to rate the average level of pain during the last 7 days on a 11 point rating scale, ranging from 0-10 (0 = "no pain" and 10 = "unbearable pain"). A lower score indicates lower severity.
Level of tenderness | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Assessed by the Fibromyalgia Impact Questionnaire Revised "level of tenderness to touch" question, asking the participants to rate the average level of tenderness to touch during the last 7 days on an 11 point rating scale, ranging from 0-10 (0 = "no tenderness" and 10 = "very tender"). A lower score indicates a lower severity.
  AND
  Assessed by measurement of pressure pain threshold, using a handheld algometer. Points measured: Right Quadriceps 15 cm proximal of apex patella and left Trapezius 10 cm from acromion. Each point is measured 3 times. Pressure pain threshold is measured in kilopascal (kPa). A higher value indicates a lower severity.
Level of fatigue | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Assessed by the Fibromyalgia Impact Questionnaire Revised "level of energy" question, asking the participants to rate the average level of energy during the last 7 days on an 11 point rating scale, ranging from 0-10 (0 = "lots of energy" and 10 = "no energy"). A lower score indicates a lower severity.
Level of sleep disturbance | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Assessed by the Fibromyalgia Impact Questionnaire Revised "quality of sleep" question asking the participants to rate the average quality of sleep during the last 7 days on an 11 point rating scale, ranging from 0-10 (0 = "awoke well rested" and 10 = "awoke very tired"). A lower score indicates a lower severity.
Level of depression | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Assessed by the Fibromyalgia Impact Questionnaire Revised "level of depression" question, asking the participants to rate the average level of depression during the last 7 days on an 11 point rating scale, ranging from 0-10 (0 = "no depression" and 10 = "very depressed"). A lower score indicates a lower severity.
Level of anxiety | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Assessed by the Fibromyalgia Impact Questionnaire Revised "level of anxiety" question, asking the participants to rate the average level of anxiety during the last 7 days on an 11 point rating scale, ranging from 0-10 (0 = "not anxious" and 10 = "very anxious"). A lower score indicates a lower severity.
Level of cognition | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Assessed by the Fibromyalgia Impact Questionnaire Revised "level of memory problems" question, asking the participants to rate the average level of memory problems during the last 7 days on an 11 point rating scale, ranging from 0-10 (0 = "good memory" and 10 = "very poor memory"). A lower score indicates a lower severity.
Level of stiffness | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Assessed by the Fibromyalgia Impact Questionnaire Revised "level of stiffness" question, asking the participants to rate the average level of stiffness during the last 7 days on an 11 point rating scale, ranging from 0-10 (0 = "no stiffness" and 10 = "severe stiffness"). A lower score indicates a lower severity.
Level of physical function | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Assessed by the physical function domain of Fibromyalgia Impact Questionnaire Revised; asking participants to rate how difficult it is to perform a list of 9 common activities over the previous 7 days on an 11 point scale, ranging from 0-10 (0 = "no difficulty" and 10 = "very difficult"). The score is characterized by the sum of the 9 scores (0-90). A lower score indicates better function.
Health-related quality of life - mobility | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) mobility domain; asking the participants to rate their mobility on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems. A lower score indicates a lower severity.
Health-related quality of life - self care | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) self care domain; asking the participants to rate their ability for self care on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems. A lower score indicates a lower severity.
Health-related quality of life - usual activities | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) usual activities domain; asking the participants to rate their ability to perform usual activities on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems. A lower score indicates a lower severity.
Health-related quality of life - pain/discomfort | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) pain/discomfort domain; asking the participants to rate their level of pain or discomfort on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems. A lower score indicates a lower severity.
Health-related quality of life - anxiety/depression | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Measured by the European Quality of Life 5 Dimensions (EQ-5D) anxiety/depression domain; asking the participants to rate their level of anxiety or depression on a 1-5 Verbal Rating Scale, a score of 1 indicating no problems, and a score of 5 indicating extreme problems. A lower score indicates a lower severity.
Health-related quality of life - global | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Measured by European Quality of Life Visual Analogue Scale (EQ-VAS), which asks the participant to rate their overall health 'today' on a 0-100 VAS. A higher score indicates a better quality of life.
Number of responders with a more than 15% improvement of pain | Number of responders after 12 weeks of treatment with LDN or LDN placebo
  A responder is defined as a subject who reports a more than 15% improvement of the primary outcome (average pain during the last 7 days) after 12 weeks of treatment with LDN or LDN-placebo. Number of responders are calculated for both the LDN group and the LDN-placebo group.
Number of responders with a more than 30% improvement of pain | Number of responders after 12 weeks of treatment with LDN or LDN placebo
  A responder is defined as a subject who reports a more than 30% improvement of the primary outcome (average pain during the last 7 days) after 12 weeks of treatment with LDN or LDN-placebo. Number of responders are calculated for both the LDN group and the LDN-placebo group.
Number of responders with a more than 50% improvement of pain | Number of responders after 12 weeks of treatment with LDN or LDN placebo
  A responder is defined as a subject who reports a more than 50% improvement of the primary outcome (average pain during the last 7 days) after 12 weeks of treatment with LDN or LDN-placebo. Number of responders are calculated for both the LDN group and the LDN-placebo group.

OTHER OUTCOMES:
Variation in pain | Change from baseline when assessed after 4, 8, and 12 weeks of treatment with LDN or LDN-placebo
  Measured using a diary of daily average pain rated on an 11 point rating scale, ranging from 0-10, during 7 days before visits at baseline, and after 8 and 12 weeks of treatment. The variation in pain is characterized by the highest score minus the lowest score. A lower score indicates a lower variation.
Muscle exhaustion | Change from baseline when assessed after 12 weeks of treatment with LDN or LDN-placebo
  Measured by an isometric muscle exhaustion test of the deltoid muscle. Measured by asking the participant to complete an isometric muscle exhaustion task by maintaining 90° shoulder abduction (dominant arm) for as long as possible with the elbow extended and the hand pronated (hand facing downwards). Task failure (test position can no longer be maintained) defines the test duration. The participants are instructed to maintain the position until they feel maximal muscle exhaustion (corresponding to a score of 10 on a 0-10 scale with 0 being "no muscle fatigue" and 10 being 'maximal muscle fatigue/exhaustion'). Surface electromyography (EMG) will be recorded from the anterior, middle and posterior deltoid muscle at 3000 Hz during the entire test. A longer duration of test is indicative of lower levels of exhaustion.
Physical fitness | Change from baseline when assessed after 12 weeks of treatment with LDN or LDN-placebo
  Measured by the 30-second chair stand test. The test starts with the subject seated on a chair with her back touching the backrest. Subjects rise to a full stand with the back straight and then sit down again to regain this cycle as many times as they can within 30 seconds. A higher number of cycles is indicative of better physical fitness.
Pain sensitivity | Change from baseline when assessed after 12 weeks of treatment with LDN or LDN-placebo
  Assessments are conducted as recommended by the 'International Association for the Study of Pain'. Computer-controlled cuff algometry is performed on lower legs in all patients to assess pressure pain threshold and pressure pain tolerance. Pressure pain threshold and pressure pain tolerance are measured in kilopascal (kPa). A higher value is indicative of lower severity.
Inhibition of pain | Change from baseline when assessed after 12 weeks of treatment with LDN or LDN-placebo
  Measured by Conditioned pain modulation (CPM). Assessments are conducted as recommended by the 'International Association for the Study of Pain'. Computer-controlled cuff algometry is performed on lower legs to assess increase in pressure pain threshold during cuff pain conditioning on the contralateral leg. Pressure pain threshold and pressure pain tolerance are measured in kilopascal (kPa). A higher value is indicative of lower severity.
Augmentation of pain | Change from baseline when assessed after 12 weeks of treatment with LDN or LDN-placebo
  Measured by Temporal Summation of Pain (TSP). Assessments are conducted as recommended by the 'International Association for the Study of Pain'. Computer-controlled cuff algometry is performed on lower legs to assess increase in pain scores to ten repeated stimulations. Pain is rated on a 0-100 Visual Analogue Scale. A lower value indicates a lower severity.

CONTACTS AND LOCATIONS:
Overall Officials: Karin D Bruun, Consultant, Principal Investigator — Odense University Hospital
Locations (1):
- Pain centre, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Due Bruun K, Christensen R, Amris K, Vaegter HB, Blichfeldt-Eckhardt MR, Bye-Moller L, Holsgaard-Larsen A, Toft P. Naltrexone 6 mg once daily versus placebo in women with fibromyalgia: a randomised, double-blind, placebo-controlled trial. Lancet Rheumatol. 2024 Jan;6(1):e31-e39. doi: 10.1016/S2665-9913(23)00278-3. Epub 2023 Dec 5. PMID 38258677
- [Derived] Bruun KD, Amris K, Vaegter HB, Blichfeldt-Eckhardt MR, Holsgaard-Larsen A, Christensen R, Toft P. Low-dose naltrexone for the treatment of fibromyalgia: protocol for a double-blind, randomized, placebo-controlled trial. Trials. 2021 Nov 15;22(1):804. doi: 10.1186/s13063-021-05776-7. PMID 34781989

DOCUMENTS (2):
  • Study Protocol (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT04270877/Prot_001.pdf
  • Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT04270877/SAP_002.pdf